CLINICAL TRIAL: NCT06508658
Title: A Phase 3, Multicenter, Randomized, Open-Label Study of Epcoritamab Plus Lenalidomide Compared to Rituximab Plus Gemcitabine and Oxaliplatin in Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Subcutaneously Injected Epcoritamab Plus Oral Lenalidomide Tablets Compared to Intravenously (IV) Infused Rituximab Plus IV Infused Gemcitabine and IV Infused Oxaliplatin in Adult Participants With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Acronym: EPCORE DLBCL-4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M22-128; 2024-510965-41 (Other: EU CT)
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Epcoritamab; Lenalidomide; Rituximab; Gemcitabine; Oxaliplatin; Diffuse Large B-Cell Lymphoma; DLBCL; Epkinly; ABBV-GMAB-3013
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Lenalidomide; Oxaliplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A: Epcoritamab Plus Lenalidomide (E-Len) (Experimental): Participants will receive E-Len for up to 12 cycles (each cycle is 28 days).
  Interventions: Drug: Epcoritamab; Drug: Lenalidomide
- Arm B: Rituximab Plus Gemcitabine and Oxaliplatin (R-GemOx) (Experimental): Participants will receive R-GemOx for up to 4 cycles (each cycle is 28 days)
  Interventions: Drug: Rituximab; Drug: Oxaliplatin; Drug: Gemcitabine
- Arm C: Epcoritamab (Experimental): Participants will receive epcoritamab for up to 12 cycles (each cycle is 28 days).
  Interventions: Drug: Epcoritamab

INTERVENTIONS:
Drug: Epcoritamab — Subcutaneous Injection
  Arms: Arm A: Epcoritamab Plus Lenalidomide (E-Len); Arm C: Epcoritamab
Drug: Rituximab — Intravenous (IV) Infusion
  Arms: Arm B: Rituximab Plus Gemcitabine and Oxaliplatin (R-GemOx)
Drug: Lenalidomide — Oral Capsule
  Arms: Arm A: Epcoritamab Plus Lenalidomide (E-Len)
Drug: Oxaliplatin — IV Infusion
  Arms: Arm B: Rituximab Plus Gemcitabine and Oxaliplatin (R-GemOx)
Drug: Gemcitabine — IV Infusion
  Arms: Arm B: Rituximab Plus Gemcitabine and Oxaliplatin (R-GemOx)

SUMMARY:
B-cell Lymphoma is an aggressive and rare cancer of a type of immune cells (a white blood cell responsible for fighting infections). This study will assess how safe and effective epcoritamab plus lenalidomide (E-Len) is compared to rituximab plus gemcitabine and oxaliplatin (R-GemOx) )in treating adult participants with relapsed or refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL). Adverse events and change in disease condition will be assessed.

Epcoritamab is an investigational drug being developed for the treatment of DLBCL. Study doctors put the participants in 1 of 3 groups, called treatment arms. Each group receives a different treatment. Around 360 adult participants with R/R DLBCL will be enrolled in approximately 165 sites across the world.

Participants in arm A will receive subcutaneous (SC) injections of epcoritamab plus oral lenalidomide capsules (E-Len) for up to 12 cycles (each cycle is 28 days). Participants in arm B will receive intravenously (IV) infused R-GemOx for up to 4 cycles (each cycle is 28 days). Participants in arm C will receive SC injections of epcoritamab for up to 12 cycles (each cycle is 28 days).

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group Performance status score of 0 to 2.
* Histologically confirmed CD20+ Diffuse Large B-Cell Lymphoma (DLBCL) and documented in the most recent and representative pathology report, inclusive of the following according to the World Health Organization (WHO) 2022 as per the protocol.
* Must have relapsed or refractory (R/R) disease and have been previously treated with at least 1 line of systemic antineoplastic therapy including anti-CD20 mAb-containing combination chemotherapy since DLBCL diagnosis.
* Participant must meet at least 1 of the following criteria:

  * Failed prior autologous stem cell transplant (ASCT), defined as relapsed after ASCT or been refractory to high-dose therapy (HDT)-ASCT.
  * Not be considered a candidate for ASCT due to age, performance status, comorbidities and/or insufficient response to prior treatment, or have refused ASCT.
  * Be ineligible for or unable to receive chimeric antigen receptor T-cell (CAR-T) meeting at least 1 of the following criteria:

    * Unable to receive CAR-T therapy due to fitness and/or comorbidity.
    * Lymphocyte apheresis failure.
    * Unwilling to receive CAR-T therapy.
    * Unable to receive CAR-T therapy due to financial, geographic, insurance, access, and/or manufacturing constraints.
    * Relapsed/progressed after having achieved at least a Partial Response (PR) or Complete Response (CR) while on prior CAR-T therapy.
* Must have measurable disease.
* Life expectancy > 3 months on standard of care treatment at the time of enrolling in the study

Exclusion Criteria:

* Current evidence of primary central nervous system (CNS) lymphoma or known CNS involvement by lymphoma including leptomeningeal disease, at screening.
* History of prior treatment with a bispecific antibody targeting CD3 and CD20 or prior treatment with rituximab plus gemcitabine and oxaliplatin (R-GemOx) or gemcitabine and oxaliplatin (GemOx).
* Documented refractoriness to lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Arm A vs Arm B: Progression-Free Survival (PFS) | Up to 4 Years
  PFS is defined as the duration from the date of randomization to the date of disease progression determined per Lugano 2014 criteria as assessed by an independent review committee (IRC), or death, whichever occurs first.

SECONDARY OUTCOMES:
Arm A vs Arm B: Percentage of Participants Who Achieve Complete response (CR) | Up to 4 Years
  CR is defined as the percentage of participants who achieve CR determined by Lugano 2014 criteria, as assessed by an IRC that is blinded to treatment arm prior to the initiation of new anti-lymphoma therapy.
Arm A vs Arm B: Overall Survival (OS) | Up to 4 Years
  OS is defined as the time from randomization to death from any cause.
Arm A vs Arm B: Percentage of Participants Who Achieve Minimal Residual Disease (MRD) Negativity Rate | Up to 4 Years
  The MRD negativity rate is defined as the percentage of participants who achieve MRD negative status prior to the initiation of new anti-lymphoma therapy.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (177):
- United States (19):
  - City of Hope National Medical Center /ID# 273338, Duarte, California
  - Valkyrie Clinical Trials /ID# 269935, Los Angeles, California
  - Desert Regional Medical Center /ID# 272437, Palm Springs, California
  - Lutheran Medical Center- Cancer Centers of Colorado /ID# 265823, Golden, Colorado
  - City Of Hope - Atlanta. /ID# 273092, Newnan, Georgia
  - Rush University Medical Center /ID# 242103, Chicago, Illinois
  - City Of Hope - Chicago /ID# 274430, Zion, Illinois
  - Northwest Cancer Center - Dyer Clinic /ID# 269787, Dyer, Indiana
  - Cancer Center of Kansas - Wichita /ID# 270117, Wichita, Kansas
  - University of Kentucky Chandler Medical Center /ID# 242087, Lexington, Kentucky
  - University of Maryland, Baltimore /ID# 242216, Baltimore, Maryland
  - Henry Ford Hospital /ID# 266446, Detroit, Michigan
  - Gulfport Memorial Hospital /ID# 268104, Gulfport, Mississippi
  - New York Medical College /ID# 265799, Valhalla, New York
  - East Carolina University - Brody School of Medicine /ID# 242227, Greenville, North Carolina
  - Thompson Cancer Survival Ctr /ID# 242149, Knoxville, Tennessee
  - Community Cancer Trials Of Utah /ID# 271715, Ogden, Utah
  - Utah Cancer Specialists - Salt Lake City /ID# 268603, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City /ID# 265329, Salt Lake City, Utah
- Argentina (3):
  - Hospital Universitario Austral /ID# 242791, Pilar, Buenos Aires
  - Fundaleu /Id# 242789, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto Alexander Fleming /ID# 263804, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
- Australia (6):
  - Canberra Hospital /ID# 265312, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital /ID# 263242, Sydney, New South Wales
  - Wollongong Hospital /ID# 244646, Wollongong, New South Wales
  - Toowoomba Hospital /ID# 263243, Toowoomba, Queensland
  - Monash Health - Monash Medical Centre /ID# 262783, Clayton, Victoria
  - Royal Perth Hospital /ID# 243790, Perth, Western Australia
- Belgium (5):
  - Universitair Ziekenhuis Brussel /ID# 242574, Jette, Brussels Capital
  - Centre Hospitalier Epicura - Hornu /ID# 265148, Boussu, Hainaut
  - Universite Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant /ID# 242565, Yvoir, Namur
  - Universitair Ziekenhuis Leuven /ID# 246671, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 264740, Roeselare, West-Vlaanderen
- Brazil (6):
  - Hospital Sao Rafael /ID# 262949, Salvador, Estado de Bahia
  - Hospital Erasto Gaertner /ID# 264049, Curitiba, Puerto Rico
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto /ID# 264045, Ribeirão Preto, São Paulo
  - Hospital Alemao Oswaldo Cruz /ID# 247418, São Paulo
  - Instituto D'Or de Pesquisa e Ensino - Regional Sao Paulo /ID# 263944, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao /ID# 242425, São Paulo
- Bulgaria (4):
  - UMHAT Sveti Georgi /ID# 242905, Plovdiv
  - UMHAT Sveti Ivan Rilski /ID# 242389, Sofia
  - SHAT Hematologic Diseases /ID# 242708, Sofia
  - UMHAT Multiprofile Hospital for Active Treatment Sveta Marina /ID# 262761, Varna
- CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 262751, Montreal, Quebec, Canada
- Chile (3):
  - Fundacion Arturo Lopez Perez /ID# 242421, Providencia, Santiago Metropolitan
  - Bradford Hill /ID# 262795, Santiago, Santiago Metropolitan
  - Clinica Alemana de Santiago /ID# 244139, Santiago
- China (26):
  - Peking University Third Hospital /ID# 242941, Beijing, Beijing Municipality
  - Fujian Province Cancer Hospital /ID# 265075, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen /ID# 264305, Xiamen, Fujian
  - Sun Yat-Sen University Cancer Center /ID# 242712, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital /ID# 242942, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University /ID# 242944, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital /Id# 242961, Harbin, Heilongjiang
  - Henan Cancer Hospital /ID# 242700, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Sc /ID# 242702, Wuhan, Hubei
  - Hubei Cancer Hospital /ID# 242963, Wuhan, Hubei
  - Jiangsu Peoples Hospital /ID# 271924, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University /ID# 242939, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University /ID# 242703, Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital /ID# 242968, Nanchang, Jiangxi
  - The First Hospital of Jilin University /ID# 242940, Changchun, Jilin
  - First Affiliated Hospital of China Medical University /ID# 242701, Shenyang, Liaoning
  - Shandong Cancer Hospital /ID# 264036, Jinan, Shandong
  - Shanghai Tongji Hospital /ID# 263952, Shanghai, Shanghai Municipality
  - Tianjin Cancer Hospital /ID# 243940, Tianjin, Tianjin Municipality
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sc /ID# 243139, Tianjin, Tianjin Municipality
  - The Affiliated Cancer Hospital of Xinjiang Medical University /ID# 242966, Ürümqi, Xinjiang
  - Yunnan Province Cancer Hospital /ID# 264057, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 242960, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine /ID# 243137, Hangzhou, Zhejiang
  - Zhejiang Cancer hospital /ID# 242711, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University /ID# 263951, Wenzhou, Zhejiang
- Croatia (6):
  - Klinicka bolnica Merkur /ID# 262619, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Sestre milosrdnice /ID# 262620, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 262617, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Osijek /ID# 262621, Osijek, County of Osijek-Baranja
  - Klinički Bolnički Centar Rijeka /ID# 266004, Rijeka, Primorje-Gorski Kotar County
  - Klinicki Bolnicki Centar (KBC) Split /ID# 262618, Split, Split-Dalmatia County
- Czechia (3):
  - Fakultní nemocnice Hradec Králové - Sokolská /ID# 264071, Hradec Králové, Hradec Kralove
  - Fakultní nemocnice v Motole /ID# 272378, Prague, Praha 5
  - Fakultni nemocnice Olomouc /ID# 262832, Olomouc
- France (7):
  - Les Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre /ID# 264068, Strasbourg, Alsace
  - CHU de CAEN - Hopital de la Cote de Nacre /ID# 243075, Caen, Calvados
  - CHRU Tours - Hopital Bretonneau /ID# 244580, Tours, Indre-et-Loire
  - Centre Hospitalier D'Avignon /ID# 243072, Avignon, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de la Cote Basque /ID# 243065, Bayonne, Pyrenees-Atlantiques
  - CHU Poitiers - La miletrie /ID# 243074, Poitiers, Vienne
  - Hopital Saint Vincent de Paul /ID# 243070, Lille
- Greece (5):
  - General Hospital of Athens Laiko /ID# 262809, Athens, Attica
  - University General Hospital Attikon /ID# 242041, Athens, Attica
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 242039, Athens
  - General University Hospital of Thessaloniki AXEPA /ID# 242038, Thessaloniki
  - Theageneio Anticancer Hospital /ID# 242036, Thessaloniki
- Hungary (7):
  - Pecsi Tudomanyegyetem Klinikai Kozpont /ID# 262924, Pécs, Baranya
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz /ID# 262901, Győr, Győr-Moson-Sopron
  - Debreceni Egyetem-Klinikai Kozpont /ID# 242451, Debrecen, Hajdú-Bihar
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz /ID# 242468, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Semmelweis Egyetem /ID# 242455, Budapest
  - Del-pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet /ID# 262923, Budapest
  - Orszagos Onkologiai Intezet /ID# 242457, Budapest
- Japan (13):
  - Fujita Health University Hospital /ID# 265968, Toyoake, Aichi-ken
  - National Hospital Organization Shikoku Cancer Center /ID# 265977, Matsuyama, Ehime
  - Kyushu University Hospital /ID# 267624, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital /ID# 264667, Fukushima, Fukushima
  - Sapporo Medical University Hospital /ID# 264928, Sapporo, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center /ID# 277258, Amagasaki, Hyōgo
  - Kagoshima University Hospital /ID# 248259, Kagoshima, Kagoshima-ken
  - Tokai University Hospital /ID# 265433, Isehara, Kanagawa
  - Shonankamakura General Hospital /ID# 277671, Kamakura, Kanagawa
  - Kansai Medical University Hospital /ID# 266018, Hirakata-shi, Osaka
  - Kindai University Hospital /ID# 265474, Sakai-shi, Osaka
  - Duplicate_Saitama Cancer Center /ID# 265277, Kitaadachi-gun, Saitama
  - University of Yamanashi Hospital /ID# 264671, Chuo-shi, Yamanashi
- Mexico (2):
  - Centro De Investigación Clinica Chapultepec /ID# 243959, Mexico City, Mexico City
  - Centro de Quimioterapia E Investigacion Sas de Cv /Id# 263293, Jalisco
- Netherlands (5):
  - Jeroen Bosch Ziekenhuis, locatie 's-Hertogenbosch /ID# 265204, 's-Hertogenbosch, North Brabant
  - OLVG - Locatie Oost /ID# 263355, Amsterdam, North Holland
  - Medisch Centrum Leeuwarden /ID# 245501, Leeuwarden, Provincie Friesland
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk /ID# 263361, Dordrecht, South Holland
  - St. Antonius Ziekenhuis /ID# 245197, Nieuwegein, Utrecht
- New Zealand (2):
  - North Shore Hospital /ID# 266060, Auckland
  - Wellington Hospital /ID# 265966, Wellington
- Poland (4):
  - Aidport sp z o.o. /ID# 262766, Poznan, Greater Poland Voivodeship
  - Pratia MCM Krakow /ID# 262882, Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Bada /ID# 263314, Warsaw, Masovian Voivodeship
  - Swietokrzyskie Centrum Onkologii Samodzielny Publiczny Zaklad Opieki Zdrowotnej /ID# 242436, Kielce, Świętokrzyskie Voivodeship
- Portugal (3):
  - Hospital da Luz /ID# 262965, Lisbon, Lisbon District
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE /ID# 262961, Porto
  - Unidade Local de Saude Sao Joao, EPE /ID# 262962, Porto
- Romania (4):
  - Fundeni Clinical Institute /ID# 266734, Bucharest, București
  - Institutul Oncologic Prof Dr. Ion Chiricuta Cluj Napoca /ID# 243753, Cluj-Napoca, Cluj
  - Institutul Regional de Oncologie /ID# 244367, Iași, Iaşi
  - Spitalul Clinic Coltea /ID# 243694, Bucharest
- Serbia (7):
  - Clinical Hospital Center Zvezdara /ID# 263059, Belgrade, Beograd
  - Institute for Oncology and Radiology of Serbia /ID# 263055, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 263057, Belgrade, Beograd
  - Clinical Hospital Center - Bežanijska Kosa /ID# 263053, Belgrade, Beograd
  - University Clinical Center Nis /ID# 263701, Niš, Nisavski Okrug
  - Institute for Oncology of Vojvodina /ID# 263052, Kamenitz, Vojvodina
  - University Clinical Center Vojvodina /ID# 264138, Novi Sad
- Singapore (3):
  - National Cancer Centre Singapore /ID# 267015, Singapore, Central Singapore
  - National University Hospital /ID# 264016, Singapore
  - Tan Tock Seng Hospital /ID# 266061, Singapore
- South Africa (5):
  - Wits Clinical Research /ID# 264656, Johannesburg, Gauteng
  - Alberts Cellular Therapy /ID# 262720, Pretoria, Gauteng
  - Capital Haematology Hospital /ID# 278955, Durban, KwaZulu-Natal
  - Constantiaberg Haematology /ID# 273041, Cape Town, Western Cape
  - Haemalife Inc. /ID# 262719, Kuils River, Western Cape
- South Korea (11):
  - Inje University - Busan Paik Hospital /ID# 262842, Busan, Busan Gwang Yeogsi
  - Dong-A University Medical Center /ID# 262841, Busan, Busan Gwang Yeogsi
  - Seoul National University Bundang Hospital /ID# 242405, Seongnam-si, Gyeonggido
  - Keimyung University Dongsan Hospital /ID# 262840, Daegu, Gyeongsangbuk-do
  - Jeonbuk National University Hospital /ID# 242958, Jeonju, Jeonrabugdo
  - Chonnam National University Hwasun Hospital /ID# 262843, Hwasun-gun, Jeonranamdo
  - Seoul National University Hospital /ID# 242407, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 242409, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 242408, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 242406, Seoul, Seoul Teugbyeolsi
  - Ulsan University Hospital /ID# 242956, Ulsan, Ulsan Gwang Yeogsi
- Taiwan (4):
  - National Taiwan University Hospital /ID# 243300, Taipei City, Taipei
  - China Medical University Hospital /ID# 242931, Taichung
  - Taichung Veterans General Hospital /ID# 242937, Taichung
  - National Cheng Kung University Hospital /ID# 243301, Tainan
- Turkey (Türkiye) (9):
  - Ankara Universitesi Fakultesi /ID# 242410, Ankara
  - Adnan Menderes University /ID# 242418, Aydin
  - Trakya University Medical Facu /ID# 242419, Edirne, Istanbul
  - Istanbul Universitesi-Cerrahpasa Cerrahpasa Tip Fakultesi /ID# 242414, Istanbul
  - Vehbi Koc vakfi Amerikan Hasta /ID# 242415, Istanbul
  - Ege University Medical Faculty /ID# 242417, Izmir
  - Ondokuz mayis University Facul /ID# 242412, Samsun
  - Istanbul Florence Nightingale Hospital /ID# 271544, Şişli
  - Karadeniz Technical University Farabi Hospital /ID# 264694, Trabzon
- United Kingdom (4):
  - Royal Cornwall Hospital /ID# 265130, Truro, Cornwall
  - NHS Lanarkshire /ID# 272332, Airdrie, North Lanarkshire
  - Nottingham City Hospital /ID# 265129, Nottingham, Nottinghamshire
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 242923, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Genmab is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-128